CLINICAL TRIAL: NCT05832307
Title: The INFLUENTIAL Trial - Inpatient FLU Vaccination Program Effectiveness: National Trial Implementing Best Practices and Learning Collaboratives
Brief Title: The INFLUENTIAL Trial- Evaluation of National Inpatient Influenza Vaccination Program
Acronym: Influential
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-1507
Record Dates: First submitted 2023-04-09; First posted 2023-04-27 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Influenza
Keywords: vaccination; influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a cluster SMART to evaluate the effectiveness of an inpatient influenza vaccination program on influenza vaccination rates during hospitalization at 12 U.S. pediatric health systems over 3 influenza vaccination seasons (Study Years 3-5). Sites will be randomized to the standardized influenza vaccination program or usual care in the first intervention season (traditional cluster RCT). Usual care and low performing sites will be re-randomized to the standardized program (intervention A) or the standardized program with an intensified implementation strategy (intervention B) in the second season. Sites will continue their programs in the third season to assess sustainability. The unit of intervention (randomization) is the site (i.e., health system).
Masking Description: Sites will be randomized 2:1 by the study statistician to intervention A vs. usual care. The randomization will be stratified by academic or academic plus community setting. This will ensure that the groups are balanced for site variables that may be correlated with the outcomes of interest. After the first intervention season, the 4 usual care sites and 6 lowest performing intervention sites (lowest change in vaccination rates from their baseline data) will be randomized 1:1 to intervention A vs. intervention B.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized inpatient influenza vaccination program (Active Comparator): Intervention A: The basic intervention is the inpatient influenza vaccination program, which will be comprised of the following core components: informatics and data analytic tools, evidenced-based education and communication, a multidisciplinary leadership team, and end-user engagement. Intervention B: The intensified intervention is the multifaceted influenza vaccination strategy (Intervention A) plus a learning collaborative with lead site facilitation during the trial period.
  Interventions: Other: Standardized inpatient influenza vaccination program
- Existing inpatient influenza vaccination practices (Active Comparator): Usual care is defined as the inpatient influenza vaccination practices that currently exist at a given site.
  Interventions: Other: Existing Influenza Vaccination Practices

INTERVENTIONS:
Other: Existing Influenza Vaccination Practices — Usual care is defined as the existing inpatient influenza vaccination practices that currently exist at a given site.
  Arms: Existing inpatient influenza vaccination practices
Other: Standardized inpatient influenza vaccination program — Intervention A: The basic intervention is the inpatient influenza vaccination program Intervention B: The intensified intervention is the multifaceted influenza vaccination strategy (Intervention A) plus a learning collaborative
  Other Names: Intervention A and B
  Arms: Standardized inpatient influenza vaccination program

SUMMARY:
This study plans to learn more about whether a stakeholder-informed, standardized inpatient vaccination program will increase influenza vaccination rates of hospitalized children across US pediatric health systems. The first part of the study is to form a multidisciplinary team of stakeholders, including parents, providers, nurses, pharmacists, informaticists, data analysts and communication experts across three sites in synthesizing a best practice implementation guide for an inpatient influenza vaccination program, which will then be piloted at these three sites.

DETAILED DESCRIPTION:
The overarching goal of this proposal is to determine whether a stakeholder-informed, standardized inpatient influenza vaccination program will increase influenza vaccination rates of hospitalized children across diverse U.S. pediatric health systems. Building upon preliminary data and experience with pediatric inpatient influenza vaccine delivery, the investigators will engage a multidisciplinary team of stakeholders in synthesizing a best practice implementation guide for an inpatient influenza vaccination program across three sites. The next phase of the study, using a novel adaptive trial design, will be to implement and test the program across 12 health systems. Finally, the investigators will evaluate the program's impact using an established dissemination and implementation framework.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months of age
* Admitted to an inpatient unit at a participating health system

Exclusion:

- Admission to critical care sites or hematology-oncology services

Exclusion Criteria:

* At least 6 months of age
* Admitted to an inpatient unit at a participating health system

Exclusion:

- Admission to critical care sites or hematology-oncology services

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22000 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Vaccine administration rate | 1 year
  proportion of influenza vaccine administrations to eligible patients during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Rao, Principal Investigator — University of Colorado, Children's Hospital Colorado
Locations (2):
- United States (2):
  - Ann and Robert Lurie's Children Hospital of Chicago, Chicago, Illinois
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT05832307/ICF_000.pdf